CLINICAL TRIAL: NCT04029506
Title: Medical Staffs Have Higher Risk for Gastrointestinal Polypoid Lesions: A Propensity Score-based Analysis
Brief Title: Medical Staff: Higher Risk for Gastrointestinal Polypoid Lesions
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Ph.D, Shandong University
Other Study IDs: 2019SDU-QILU-G100
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: the Incidence of Gastrointestinal Diseases Diagnosed by Endoscopy in Physicians and General Population

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- medical staff group: medical staff in Qilu Hospital who recieveing endoscopy for physical examination
- general population group: general population who recieveing endoscopy for physical examination in Qilu Hospital

INTERVENTIONS:
Other:  — this is an obsevational study which needs no interventions
  Groups: medical staff group

SUMMARY:
This is a single center, retrospective, propensity score-matched analyzed study. Patients who underwent gastroscopy and colonoscopy for physical examination in Qilu Hospital of Shandong University, China, from January 2017 to September 2018, were retrospectively reviewed to compare the incidence of gastrointestinal diseases diagnosed by endoscopy between physicians and general population.

DETAILED DESCRIPTION:
This is a single center, retrospective, propensity score-matched analyzed study. Patients who underwent gastroscopy and colonoscopy for physical examination in Qilu Hospital of Shandong University, China, from January 2017 to September 2018, were retrospectively reviewed.To compare the incidence of gastrointestinal diseases diagnosed by endoscopy between physicians and general population.

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent gastroscopy and colonoscopy for physical examination in Qilu Hospital from January 2017 to September 2018

Exclusion Criteria:

- Subjects who had a history of gastrointestinal surgery or subjects who did not finish the endoscopic examination were excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent gastroscopy and colonoscopy for physical examination in Qilu Hospital of Shandong University, China, from January 2017 to September 2018, were retrospectively reviewed. Subjects who had a history of gastrointestinal surgery or subjects who did not finish the endoscopic examination were excluded. All selected subjects were age- and sex- matched to form two groups: Group 1, medical staff from Qilu Hospital, and Group 2, general population.
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
the incidence of gastrointestinal diseases diagnosed by endoscopy between physicians and general population. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China